CLINICAL TRIAL: NCT06778707
Title: External Oblique Intercostal Block vs Subcostal Transversus Abdominis Plane Block for Adequate Analgesia in Open Nephrectomy
Brief Title: External Oblique Intercostal Block vs Subcostal Transversus Abdominis Plane Block in Open Nephrectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Wahed Ali, Lecturer at anesthesia & surgical ICU & Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR998/12/24
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Analgesia , Open Renal Surgeries
Keywords: External Oblique Intercostal Block; Subcostal Transversus Abdominis Plane Block
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blinded prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group E (Active Comparator): This group of patients will receive external oblique intercostal block in supine position. A high-frequency linear transducer will be placed in sagittal plane between the midclavicular and anterior axillary line at the level of the 6 to 8th rib. The pointing mark of the probe will be directed cranially and may be slightly tilted medially for better identification of external oblique muscle and intercostal muscles.
  After sterilization of skin and through the in-plane technique directing from cranial to caudal, a needle will be used to pierce the skin, subcutaneous tissue then external oblique muscle to hydrodissect the fascial plane between external oblique muscle and intercostal muscles with 25 ml bupivacaine 0.25 % and 4 mg dexamethasone added to it.
  Interventions: Procedure: External Oblique Intercostal Block
- group T (Active Comparator): Subcostal transversus abdominis plane block will be applied to this group and patients will be supine. A high-frequency linear transducer will be placed directly below and along costal margin. After sterilization of skin, with in-plane technique and from lateral to medial, a needle will be used to pierce the skin, subcutaneous tissue then rectus muscle and 25 ml of 0.25 % bupivacaine with 4 mg dexamethasone will be injected between rectus muscle and transversus abdominis muscle.
  Interventions: Procedure: Subcostal Transversus Abdominis Plane Block

INTERVENTIONS:
Procedure: External Oblique Intercostal Block — In group E, a needle will be used to pierce the skin, subcutaneous tissue then external oblique muscle to hydrodissect the fascial plane between external oblique muscle and intercostal muscles with 25 ml bupivacaine 0.25 % and 4 mg dexamethasone added to it.
  Arms: group E
Procedure: Subcostal Transversus Abdominis Plane Block — In group T, a needle will be used to pierce the skin, subcutaneous tissue then rectus muscle and 25 ml of 0.25 % bupivacaine with 4 mg dexamethasone will be injected between rectus muscle and transversus abdominis muscle.
  Arms: group T

SUMMARY:
The aim of the study is to compare the analgesic efficacy of external oblique intercostal block vs subcostal transversus abdominis plane block in patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
This randomized controlled double blinded study will be done on 80 patients (40 in each group), patients will be randomly classified by computer generated numbers. Through a sealed opaque envelope technique, a blinded nurse who will not participate in the study or data collection, will read the number contained in the envelope and make group assignments.

All patients will be seen in the anesthesia clinic, optimization of general condition and all required investigations will be done before surgery. Patients will be premedicated with 1.5 mg midazolam and 4 mg granisetron. Basic monitoring will be applied to the patients such as Pulse oximetry (SPO2), Non-invasive blood pressure (NIBP), Electrocardiogram (ECG), Capnogram and temperature probe.

After adequate preoxygenation, induction of general anesthesia will be done through wide bore cannula using 1 mic/kg fentanyl, 1-2 mg/kg titration of propofol, 0.5mg/kg atracurium. Patients were mechanically ventilated using volume-controlled ventilation (VCV) with adjustment of end tidal carbon dioxide (ETCO2) to be 32-35 mmHg, 50% inspired oxygen in air and sevoflurane concentration to be 1MAC. The patients will receive either block before skin incision that will be done 20 minutes after the block. 0.5 mic/kg fentanyl will be injected when heart rate or blood pressure increases more than 20% of baseline. By the end of the surgery, 1gm paracetamol will be administered with fully reversal of muscle relaxants at the end of the surgery.

Group E This group of patients will receive external oblique intercostal block in supine position. A high-frequency linear transducer will be placed in sagittal plane between the midclavicular and anterior axillary line at the level of the 6 to 8th rib. The pointing mark of the probe will be directed cranially and may be slightly tilted medially for better identification of external oblique muscle and intercostal muscles.

After sterilization of skin and through the in-plane technique directing from cranial to caudal, a needle will be used to pierce the skin, subcutaneous tissue then external oblique muscle to hydrodissect the fascial plane between external oblique muscle and intercostal muscles with 25 ml bupivacaine 0.25 % and 4 mg dexamethasone added to it.

Group T Subcostal transversus abdominis plane block will be applied to this group and patients will be supine. A high-frequency linear transducer will be placed directly below and along costal margin. After sterilization of skin, with in-plane technique and from lateral to medial, a needle will be used to pierce the skin, subcutaneous tissue then rectus muscle and 25 ml of 0.25 % bupivacaine with 4 mg dexamethasone will be injected between rectus muscle and transversus abdominis muscle.

After extubation, the patients will be transferred to PACU (Post-Anesthesia Care Unit) for monitoring. Numerical rating scale (NRS) will be used for pain assessment while 0 is no pain and 10 is severe agonizing pain. Patients will be given a rescue analgesia of 0.05 mg / kg morphine if NRS ≥ 4 and repeated if needed after 20 minutes. 1 gm paracetamol every 8 h and 30 mg ketorolac (if not contraindicated) every 12 h will be given regularly.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be included in the study age from 21 to 60 years, both male and female, with American Society of Anesthesiologists (ASA) Physical Status Classification System I-III.

Exclusion Criteria:

* Any patient refuses to participate, has bleeding or coagulation disorders, hepatic dysfunction, psychiatric diseases, on chronic opioid use, with history of allergy to local anesthetics and has infection at the needle entry point will be excluded.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption in the first postoperative 24 hour | first postoperative 24 hour
  Total morphine consumption in the first postoperative 24 hour

SECONDARY OUTCOMES:
NRS when patient reach recovery room and at 2 hour, 6 hour, 12 hour, 18 hour and 24 hour | when patient reach recovery room and at 2 hour, 6 hour, 12 hour, 18 hour and 24 hour
  NRS when patient reach recovery room and at 2 hour, 6 hour, 12 hour, 18 hour and 24 hour
Total intraoperative fentanyl consumption with exclusion of fentanyl used in induction | intraoperative
  Total intraoperative fentanyl consumption with exclusion of fentanyl used in induction

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelwahed, lecturer, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing abstract and final paper on a medical journal
Supporting Information: Study Protocol
Time Frame: data will be available after finishing the study within one year
Access Criteria: google scholar

REFERENCES:
- [Background] 1.Bansal P, Sultania N, Mittal T. External oblique intercostal block in open nephrectomy patients-A zenith in analgesia for anterolateral upper abdominal surgeries: A case series. Asian Journal of Medical Sciences. 2024;15(2):264-8.
- See also: https://ajmsjournal.info/index.php/AJMS/article/view/382?articlesBySimilarityPage=15 — https://ajmsjournal.info/index.php/AJMS/article/view/382?articlesBySimilarityPage=15